CLINICAL TRIAL: NCT01028911
Title: A Phase 1, Double-Blind, Placebo-Controlled, Sponsor-Open, Randomized, Multiple Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PF-03654746 in Mild to Moderate Alzheimer's Disease Patients on Stable Donepezil Therapy
Brief Title: A Study to Evaluate the Safety, Tolerability, and Blood Levels of PF-03654746 in Subjects With Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study terminated 27Apr2010 due to slow recruitment and the need to use the existing information to determine dosing for another study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A8801016
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Alzheimer's Disease
Keywords: Phase 1 Alzheimer's disease Safety Tolerability Pharmacokinetics
MeSH Terms: conditions — Alzheimer Disease | interventions — N-ethyl-3-fluoro-3-(3-fluoro-4-(pyrrolidinylmethyl)phenyl)cyclobutanecarboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-03654746 (Experimental)
  Interventions: Drug: PF-03654746
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-03654746 — PF-03654746 capsule of 0.25 mg, 0.5 mg, and 1.0 mg strength. Drug is dosed orally once a day. Forced titration dosing for the first 15 days of the study being at 0.25 mg for 5 days, then 0.5 mg for days 6-10, then 1.0 mg for days 11-15. Flexible dosing for the next 15 days depending on tolerability and safety assessments done by the investigator.
  Arms: PF-03654746
Drug: Placebo — Matching placebo capsules to PF-03654746 with strengths of 0.25 mg, 0.5 mg, and 1.0 mg.
  Drug is dosed orally once a day. Forced titration dosing for the first 15 days of the study being at 0.25 mg for 5 days, then 0.5 mg for days 6-10, then 1.0 mg for days 11-15. Flexible dosing for the next 15 days depending on tolerability and safety assessments done by the investigator.
  Arms: Placebo

SUMMARY:
This is a study to evaluate the safety, tolerability and blood levels of PF-03654746 in subjects will mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's disease
* Mini Mental State Examination score 18-26 inclusive
* Aged 55-85

Exclusion Criteria:

* Dementia other than Alzheimer's disease
* Clinically significant cardiovascular disease in the past 6 months prior to screening
* Creatinine clearance <30 mL/min

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Wichita, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8801016&StudyName=A%20Study%20to%20Evaluate%20the%20Safety%2C%20Tolerability%2C%20and%20Blood%20Levels%20of%20PF-03654746%20in%20Subjects%20with%20Mild%20to%20Moderate%20Alzheimer%27s%20Diseas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were on a stable dose of donepezil (Aricept) 10 milligram (mg) once daily for at least 30 days before screening and on stable morning dosing at least 14 days before Day 0 were enrolled in this study.
Groups:
- PF-03654746 and Donepezil: PF-03654746 0.25 milligram (mg) powder in capsule orally once daily on Day 1 to 5, followed by PF-03654746 0.5 mg powder in capsule orally once daily on Day 6 to 10 and PF-03654746 1 mg powder in capsule orally once daily on Day 11 to 15 during the forced titration phase. PF-03654746 0.5 mg to 2 mg powder in capsule orally once daily, based on investigator's discretion and tolerability, on Day 16 to 30 during the flexible titration phase. Background donepezil (Aricept) 10 mg tablet orally once daily throughout the study.
- Placebo and Donepezil: Placebo matched to PF-03654746 powder in capsule once daily on Day 1 to 30 along with background donepezil (Aricept) 10 mg tablet orally once daily throughout the study.
Period: Overall Study
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Started | 7 | 2
Completed | 7 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Customized [Number; unit: participants]
  45 to 64 years | 1 | 0 | 1
  Greater than or equal to (>=) 65 years | 6 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Criteria for potential clinical concern in vital signs: supine and standing systolic blood pressure (SBP) less than (<) 90 millimeter of mercury (mmHg), supine and standing diastolic BP (DBP) <50 mmHg, supine pulse rate <40 beats per minute (bpm) or >120 bpm, standing pulse rate <40 bpm or >140 bpm. Maximum increase or decrease from baseline in supine (Su) and standing (St) SBP >=30 mmHg and maximum increase or decrease from baseline in supine and standing DBP >=20 mmHg.
Time Frame: Baseline up to 7 to 10 days after last dose
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
participants
  Supine SBP <90 mmHg | 0 | 0
  Standing SBP <90 mmHg | 0 | 0
  Supine DBP <50 mmHg | 0 | 0
  Standing DBP <50 mmHg | 0 | 0
  Supine pulse rate <40 bpm | 0 | 0
  Supine pulse rate >120 bpm | 0 | 0
  Standing pulse rate <40 bpm | 0 | 0
  Standing pulse rate >140 bpm | 0 | 0
  Su SBP: Maximum increase from baseline >=30 mmHg | 3 | 0
  St SBP: Maximum increase from baseline >=30 mmHg | 1 | 0
  Su DBP: Maximum increase from baseline >=20 mmHg | 2 | 0
  St DBP: Maximum increase from baseline >=20 mmHg | 1 | 0
  Su SBP: Maximum decrease from baseline >=30 mmHg | 0 | 1
  St SBP: Maximum decrease from baseline >=30 mmHg | 0 | 0
  Su DBP: Maximum decrease from baseline >=20 mmHg | 0 | 0
  St DBP: Maximum decrease from baseline >=20 mmHg | 1 | 1

2. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for potential clinical concern in ECG parameters: maximum PR interval of >=300 milliseconds (msec), maximum QRS interval >=200 msec, maximum fridericia's corrected QT (QTcF) interval >=500 msec, PR interval or QRS interval increase from baseline >=25 percent (%) or 50 percent (%), QTCF interval increase from baseline 30 to 60 msec or >=60 msec.
Time Frame: Baseline up to 7 to 10 days after last dose
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
participants
  Maximum PR interval >=300 msec | 0 | 0
  Maximum QRS Complex >=200 msec | 0 | 0
  Maximum QTCF interval >=500 msec | 1 | 0
  PR interval increase from baseline >=25/50 % | 0 | 0
  QRS complex increase from baseline >=25/50 % | 0 | 0
  QTCF interval increase from baseline 30 to 60 msec | 2 | 0
  QTCF interval increase from baseline >=60 msec | 1 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities
Description: Criteria for laboratory tests abnormalities included: hemoglobin, hematocrit and red blood cells (< 0.8*lower limit of normal[LLN]); leucocytes (<0.6/>1.5*upper limit of normal [ULN]); platelets (<0.5*LLN/>1.75*ULN); neutrophils, lymphocytes (<0.8*LLN/>1.2*ULN); eosinophils, basophils, monocytes (>1.2*ULN); total bilirubin (>1.5*ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (>3*ULN), total protein, albumin (<0.8*LLN/>1.2*ULN); creatinine, urea (>1.3*ULN); glucose (<0.6*LLN/>1.5*ULN); uric acid (>1.2*ULN); sodium, potassium, chloride, calcium, bicarbonate (<0.9*LLN/>1.1*ULN); urine red blood cells (RBCs), urine white blood cells (WBCs), urine epithelial cells (>=6 high-powered field), urine bacteria >20 high-powered field; qualitative urine glucose, ketones, protein values >=1 in urine dipstick test. Total number of participants with any laboratory abnormalities was reported.
Time Frame: Baseline up to 7 to 10 days after last dose
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
participants | 7 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination
Description: Physical examination included examination of the skin, eyes, ears, throat, neck, and cardiac, respiratory, gastrointestinal and musculoskeletal systems. The examination assessed the participants for any potential changes in physical status, as determined by the investigator. Any untoward findings identified on physical exams conducted after the administration of the first dose of study medication was captured as an adverse event.
Time Frame: Baseline up to 7 to 10 days after last dose
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
participants | 0 | 0

5. Primary Outcome: Medical Outcomes Study - Sleep Scale (MOS-SS) Score at Baseline
Description: Participant-rated 12-item questionnaire to assess sleep quality and quantity. The items contribute to each scale and are averaged to create the 7 subscale scores: sleep disturbance, snoring, awaken short of breath (ASoB) or with a headache, somnolence, sleep adequacy, sleep quantity (range 0 to 24) and optimal sleep (yes: 1, no: 0), and overall sleep problem index (SPI) I and II. Except for sleep quantity and optimal sleep, scores are transformed (actual raw score minus lowest possible score divided by possible raw score range* 100); total score range: 0 to 100; higher score = greater intensity of attribute. Except for sleep quantity, sleep adequacy and optimal sleep, higher scores=greater impairment. Scales with at least one item answered was used to generate a scale score.
Time Frame: Baseline
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale
  Sleep disturbance | 23.76 (21.57) | 15.65 (22.13)
  Somnolence | 30.49 (18.40) | 16.70 (14.14)
  Sleep adequacy | 65.71 (32.07) | 85.00 (21.21)
  Snore | 45.71 (37.80) | 20.00 (28.28)
  Awaken short of breath or with headache | 8.57 (15.74) | 0.00 (0.00)
  Quantity of sleep | 7.86 (0.90) | 10.50 (2.12)
  Optimal sleep | 0.71 (0.49) | 0.00 (0.00)
  Sleep problem index I | 23.81 (17.70) | 10.00 (14.14)
  Sleep problem index II | 24.21 (15.81) | 14.70 (17.68)

6. Primary Outcome: Medical Outcomes Study - Sleep Scale (MOS-SS) Score at Day 5
Description: as for outcome 5
Time Frame: Day 5
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale
  Sleep disturbance | 25.01 (19.56) | 15.65 (22.13)
  Somnolence | 28.57 (26.87) | 16.70 (14.14)
  Sleep adequacy | 65.71 (22.25) | 90.00 (14.14)
  Snore | 28.57 (30.24) | 20.00 (28.28)
  Awaken short of breath or with headache | 8.57 (22.68) | 0.00 (0.00)
  Quantity of sleep | 7.57 (0.98) | 9.50 (0.71)
  Optimal sleep | 0.71 (0.49) | 0.00 (0.00)
  Sleep problem index I | 21.89 (14.25) | 8.35 (11.81)
  Sleep problem index II | 24.76 (14.64) | 13.60 (16.12)

7. Primary Outcome: Medical Outcomes Study - Sleep Scale (MOS-SS) Score at Day 10
Description: as for outcome 5
Time Frame: Day 10
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale
  Sleep disturbance | 27.69 (27.86) | 13.15 (18.60)
  Somnolence | 29.53 (31.46) | 16.70 (14.14)
  Sleep adequacy | 67.14 (29.28) | 90.00 (14.14)
  Snore | 34.29 (35.99) | 20.00 (28.28)
  Awaken short of breath or with headache | 14.29 (37.80) | 0.00 (0.00)
  Quantity of sleep | 7.43 (1.13) | 9.50 (0.71)
  Optimal sleep | 0.57 (0.53) | 0.00 (0.00)
  Sleep problem index I | 26.19 (20.14) | 8.35 (11.81)
  Sleep problem index II | 26.90 (19.49) | 12.50 (14.57)

8. Primary Outcome: Medical Outcomes Study - Sleep Scale (MOS-SS) Score at Day 15
Description: as for outcome 5
Time Frame: Day 15
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale
  Sleep disturbance | 28.76 (11.58) | 13.15 (18.60)
  Somnolence | 28.57 (20.27) | 16.70 (14.14)
  Sleep adequacy | 64.29 (31.01) | 90.00 (14.14)
  Snore | 40.00 (41.63) | 20.00 (28.28)
  Awaken short of breath or with headache | 5.71 (15.12) | 0.00 (0.00)
  Quantity of sleep | 7.29 (0.95) | 9.50 (0.71)
  Optimal sleep | 0.71 (0.49) | 0.00 (0.00)
  Sleep problem index I | 28.10 (16.55) | 8.35 (11.81)
  Sleep problem index II | 26.74 (15.20) | 12.50 (14.57)

9. Primary Outcome: Medical Outcomes Study - Sleep Scale (MOS-SS) Score at Day 20
Description: as for outcome 5
Time Frame: Day 20
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale
  Sleep disturbance | 23.57 (22.07) | 5.65 (7.99)
  Somnolence | 37.14 (30.75) | 10.00 (14.14)
  Sleep adequacy | 61.43 (26.10) | 95.00 (7.07)
  Snore | 42.86 (43.86) | 10.00 (14.14)
  Awaken short of breath or with headache | 8.57 (15.74) | 0.00 (0.00)
  Quantity of sleep | 7.00 (1.41) | 9.50 (0.71)
  Optimal sleep | 0.43 (0.53) | 0.00 (0.00)
  Sleep problem index I | 26.19 (18.11) | 3.35 (4.74)
  Sleep problem index II | 26.67 (18.20) | 5.85 (8.27)

10. Primary Outcome: Medical Outcomes Study - Sleep Scale (MOS-SS) Score at Day 25
Description: as for outcome 5
Time Frame: Day 25
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale
  Sleep disturbance | 23.76 (21.18) | 3.15 (4.45)
  Somnolence | 36.19 (28.24) | 6.65 (9.40)
  Sleep adequacy | 72.86 (22.15) | 95.00 (7.07)
  Snore | 45.71 (47.21) | 10.00 (14.14)
  Awaken short of breath or with headache | 5.71 (15.12) | 0.00 (0.00)
  Quantity of sleep | 7.71 (0.95) | 9.50 (0.71)
  Optimal sleep | 0.71 (0.49) | 0.00 (0.00)
  Sleep problem index I | 22.37 (16.86) | 1.65 (2.33)
  Sleep problem index II | 23.89 (16.04) | 3.60 (5.09)

11. Primary Outcome: Medical Outcomes Study - Sleep Scale (MOS-SS) Score at Day 30
Description: as for outcome 5
Time Frame: Day 30
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale
  Sleep disturbance | 23.04 (21.99) | 3.15 (4.45)
  Somnolence | 37.16 (24.62) | 6.65 (9.40)
  Sleep adequacy | 72.86 (22.15) | 95.00 (7.07)
  Snore | 42.86 (43.86) | 10.00 (14.14)
  Awaken short of breath or with headache | 5.71 (15.12) | 0.00 (0.00)
  Quantity of sleep | 7.86 (1.07) | 9.50 (0.71)
  Optimal sleep | 0.57 (0.53) | 0.00 (0.00)
  Sleep problem index I | 21.90 (17.52) | 1.65 (2.33)
  Sleep problem index II | 23.26 (16.21) | 3.60 (5.09)

12. Primary Outcome: Medical Outcomes Study - Sleep Scale (MOS-SS) Score at Follow-up
Description: as for outcome 5
Time Frame: Follow-up (7 to 10 days after last dose)
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale
  Sleep disturbance | 16.44 (17.07) | 3.15 (4.45)
  Somnolence | 32.39 (27.62) | 6.65 (9.40)
  Sleep adequacy | 72.86 (23.60) | 95.00 (7.07)
  Snore | 42.86 (43.86) | 10.00 (14.14)
  Awaken short of breath or with headache | 5.71 (15.12) | 0.00 (0.00)
  Quantity of sleep | 8.14 (0.69) | 9.50 (0.71)
  Optimal sleep | 0.71 (0.49) | 0.00 (0.00)
  Sleep problem index I | 17.61 (15.25) | 1.65 (2.33)
  Sleep problem index II | 19.67 (14.12) | 3.60 (5.09)

13. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score at Day 5
Description: NPI: 12-domain caregiver assessment of behavioral disturbances occurring in dementia: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, appetite/eating, night-time behavior. Severity (1=Mild to 3=Severe), frequency (1=occasionally to 4=very frequently) scales recorded for each domain; frequency*severity=each domain score (range 0-12). Total score=sum of each domain score (range 0-144); higher score=greater behavioral disturbances; negative change score from baseline=improvement.
Time Frame: Baseline, Day 5
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale
  Baseline | 4.1 (6.09) | 3.0 (4.24)
  Change at Day 5 | -1.9 (5.64) | -1.0 (1.41)

14. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score at Day 10
Description: as for outcome 13
Time Frame: Baseline, Day 10
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | -1.7 (4.75) | -1.0 (1.41)

15. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score at Day 15
Description: as for outcome 13
Time Frame: Baseline, Day 15
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | -2.6 (4.39) | -1.0 (1.41)

16. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score at Day 20
Description: as for outcome 13
Time Frame: Baseline, Day 20
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | -2.7 (5.71) | 0.0 (0.00)

17. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score at Day 25
Description: as for outcome 13
Time Frame: Baseline, Day 25
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | -2.6 (4.39) | 0.0 (0.00)

18. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score at Day 30
Description: as for outcome 13
Time Frame: Baseline, Day 30
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | -1.4 (5.22) | 0.0 (0.00)

19. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score at Follow-up
Description: as for outcome 13
Time Frame: Baseline, Follow-up (7 to 10 days after last dose)
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | -2.6 (4.39) | 1.5 (2.12)

20. Primary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score at Day 5
Description: MMSE measured general cognitive functioning: orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two intersecting polygons. Total score derived from sub-scores; total ranged from 0 to 30, higher score indicates better cognitive state.
Time Frame: Baseline, Day 5
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale
  Baseline | 24.6 (1.51) | 24.0 (0.00)
  Change at Day 5 | -0.7 (2.29) | 3.0 (0.00)

21. Primary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score at Day 10
Description: as for outcome 20
Time Frame: Baseline, Day 10
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | 0.1 (2.34) | 3.0 (0.00)

22. Primary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score at Day 15
Description: as for outcome 20
Time Frame: Baseline, Day 15
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | 1.3 (1.80) | 2.5 (0.71)

23. Primary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score at Day 20
Description: as for outcome 20
Time Frame: Baseline, Day 20
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | 0.4 (2.94) | 4.0 (0.00)

24. Primary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score at Day 25
Description: as for outcome 20
Time Frame: Baseline, Day 25
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | 1.0 (2.08) | 3.5 (0.71)

25. Primary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score at Day 30
Description: as for outcome 20
Time Frame: Baseline, Day 30
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | 0.6 (2.37) | 3.0 (2.83)

26. Primary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score at Follow-up
Description: as for outcome 20
Time Frame: Baseline, Follow-up (7 to 10 days after last dose)
Population: Safety population included all participants who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
units on a scale | 0.7 (1.60) | 3.0 (4.24)

27. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for PF-03654746
Time Frame: 0 hour (pre-dose), 0.5, 1, 3, 8 and 12 hours post-dose on Day 30
Population: Pharmacokinetic (PK) parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest during the study.
Measure: Geometric Mean (Standard Deviation); unit: nanogram hour per milliliter (ng*hr/mL)
Arm/Group | PF-03654746 and Donepezil
Number analyzed (Participants) | 7
nanogram hour per milliliter (ng*hr/mL) | 118.6 (35.687)

28. Secondary Outcome: Maximum Serum Concentration (Cmax) for PF-03654746
Time Frame: 0 hour (pre-dose), 0.5, 1, 3, 8 and 12 hours post-dose on Day 30
Population: PK parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest during the study.
Measure: Geometric Mean (Standard Deviation); unit: nanogran per millileter (ng/mL)
Arm/Group | PF-03654746 and Donepezil
Number analyzed (Participants) | 7
nanogran per millileter (ng/mL) | 9.430 (2.7317)

29. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) for PF-03654746
Time Frame: 0 hour (pre-dose), 0.5, 1, 3, 8 and 12 hours post-dose on Day 30
Population: as for outcome 28
Measure: Median (Full Range); unit: hours
Arm/Group | PF-03654746 and Donepezil
Number analyzed (Participants) | 7
hours | 3.00 [1.00 to 3.00]

30. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for Donepezil
Time Frame: 0 hour (pre-dose), 0.5, 1, 3, 8, 12 hours post-dose on Day 0, Day 30
Population: as for outcome 28
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
ng*hr/mL
  Day 0 | 881.6 (282.03) | 1109 (176.07)
  Day 30 | 1035 (364.62) | 1013 (91.217)
Statistical Analysis 1: Comparison: PF-03654746 and Donepezil vs Placebo and Donepezil; Day 30: Natural log transformed AUCtau of donepezil was analyzed using a mixed effect model with sequence, day and treatment as fixed effects and participant within sequence as a random effect.The adjusted mean differences and 90% confidence intervals for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios. Values were back-transformed from the log scale; Test type: Superiority or Other; Adjusted Geometric Means Ratio = 128.40, 90% CI 2-sided [75.90 to 217.21]

31. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Donepezil
Time Frame: 0 hour (pre-dose), 0.5, 1, 3, 8, 12 hours post-dose on Day 0, Day 30
Population: as for outcome 28
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
ng/mL
  Day 0 | 45.47 (12.847) | 53.89 (10.465)
  Day 30 | 50.28 (14.864) | 49.73 (1.7678)
Statistical Analysis 1: Comparison: PF-03654746 and Donepezil vs Placebo and Donepezil; [analysis description as in outcome 30, analysis 1]; Test type: Superiority or Other; Adjusted Geometric Means Ratio = 119.82, 90% CI 2-sided [75.90 to 189.16]

32. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Donepezil
Time Frame: 0 hour (pre-dose), 0.5, 1, 3, 8, 12 hours post-dose on Day 0, Day 30
Population: as for outcome 28
Measure: Median (Full Range); unit: hours
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Number analyzed (Participants) | 7 | 2
hours
  Day 0 | 2.98 [0.967 to 3.00] | 2.99 [2.98 to 3.00]
  Day 30 | 3.00 [2.98 to 12.0] | 2.98 [2.98 to 2.98]

ADVERSE EVENTS:
Arm/Group | PF-03654746 and Donepezil | Placebo and Donepezil
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 5/7 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03654746 and Donepezil (N=7) | Placebo and Donepezil (N=2)
Headache (Nervous system disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0
Hypnagogic hallucination (Psychiatric disorders) | 1 | 0
Illusion (Psychiatric disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to slow recruitment and the need to use the existing information to determine dosing for another study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.